CLINICAL TRIAL: NCT00945295
Title: Open-label, Parallel Study to Determine the Efficacy and Safety of Botulinum Neurotoxin A Paired With Rehabilitation Therapy vs. Botulinum Neurotoxin A Alone for the Treatment of Post-stroke Upper Limb Spasticity
Brief Title: Efficacy and Safety Study of Botulinum Neurotoxin A With Rehabilitation Versus Botulinum Neurotoxin A Alone in Treatment of Post-stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JoAnn Harnar (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, JoAnn Harnar, Research Nurse, Biomedical Research Institute of New Mexico
Organization: Biomedical Research Institute of New Mexico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Allergan-100808
Record Dates: First submitted 2009-03-30; First posted 2009-07-24 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-08

CONDITIONS: Upper Limb Spasticity
Keywords: Cerebrovascular Accident/Rehabilitation; Muscle Spasticity; Botulinum Neurotoxin Type A; Post-stroke focal upper limb spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort #1 (Active Comparator): Cohort 1 will receive BoNT-A plus rehabilitation therapy for the duration of the study (for up to 2 injections of BoNT-A).
  Interventions: Drug: Botulinum toxin type A, BoNT-A; Other: Rehabilitation Therapy
- Cohort #2 (Active Comparator): Cohort 2 will receive BoNT-A alone
  Interventions: Drug: Botulinum toxin type A, BoNT-A

INTERVENTIONS:
Drug: Botulinum toxin type A, BoNT-A — Participants will receive IM injections of BoNT-A between 200 and 400 Units with the total dose not to exceed 6 U / kg. The primary targets for BoNT-A injection are the wrist and finger flexor muscles (flexor carpi radialis, flexor carpi ulnaris, flexor digitorum profundus, flexor digitorum superficialis).
Other: Rehabilitation Therapy — Rehabilitation therapy
  Arms: Cohort #1

SUMMARY:
The purpose of this study is to determine if a combination of botulinum neurotoxin A and rehabilitation therapy is better than botulinum neurotoxin A alone for improvement in function based on the Fugl-Meyer and other validated measures.

Hypothesis: The combination of botulinum neurotoxin A and rehabilitation therapy will produce better functional improvement than botulinum neurotoxin A alone in post-stroke upper limb spasticity measured by the Fugl-Meyer Assessment of Sensorimotor Recovery after Stroke.

DETAILED DESCRIPTION:
This trial is a multi-center, parallel design comparing open label BoNT-A paired with rehabilitation therapy (OT) versus BoNT-A alone in patients diagnosed with post-stroke focal upper limb spasticity. Cohort 1 will receive BoNT-A plus rehabilitation therapy for the duration of the study (for up to 2 injections of BoNT-A) while Cohort 2 will receive BoNT-A alone. The injection protocol will closely follow the design of the Allergan 191622-056 study with the inclusion of rehabilitation therapy intervention. Those randomized to BoNT-A alone will not be able to start any new therapy or exercise therapy while in the study. Two types of patients will be recruited for the study, those naïve to BoNT-A and those who have received BoNT-A for treatment of their spasticity. Given that BoNT-A has temporary effects, the second group of patients is not expected to react differently that patients naïve to the intervention. The sites will contact patients previously enrolled in the 191622-008, 025 and 056 protocols to determine if they are eligible for involvement in the BoNT-A / rehabilitation study. In addition, the sites will recruit from the local community patients who have and have not received BoNT-A treatment for their spasticity by placing a notice in the stroke club newsletters, contacting local physician and rehabilitation offices, and posting fliers in area hospitals. Patients will be screened for eligibility during an interview with a study team member. Eligible patients will complete the informed consent process, sign a consent form, HIPPA. A blinded study physician will perform a physical examination and focal exam of the affected limb obtaining Modified Ashworth Scale scores for the elbow, wrist, finger, and thumb. Following the baseline visit, appointments will be scheduled for the next visit (Study Visit 1 {Week 0}, injection of BoNT-A. Prior to injection,, patients will be evaluated by a Therapist, blinded to treatment who will do the Functional Independence Measure (FIM) and the Fugl-Meyer Assessment of Sensorimotor Recovery after Stroke (Upper Extremity subsection). Participants will receive IM injections of BoNT-A between 200 and 400 Units with the total dose not to exceed 6 U / kg. The primary targets for BoNT-A injection are the wrist and finger flexor muscles (flexor carpi radialis, flexor carpi ulnaris, flexor digitorum profundus, flexor digitorum superficialis). Additional target muscles include biceps, brachioradialis, brachialis, pronator quadratus, pronator teres, flexor pollicis brevis / opponens, adductor pollicis, flexor pollicis longus, and lumbricales / interossei. The goal of the injections is to reduce spasticity causing such events as flexed elbow, pronated forearm, flexed wrist, thumb in palm, clenched fist, and hand deformity. It is not necessary to administer the same dose or inject the same muscles at each injection visit. The treatment should be guided by the spasticity measured and the clinical judgment of the Investigator. All injections will be performed with the assistance of EMG guidance for muscle localization. Randomization to either BoNT-A + rehab or BoNT-A alone will occur after the first injection. Randomization schedule will be determined by sequential lettered sealed envelopes sent to each site, generated by the independent analyst.

Participants assigned to Cohort 1 (determined by a randomization scheme) will also be scheduled for weekly therapy appointments to begin within 2 weeks of injection. An attempt will be made to have all study patients seen by the same therapists at each site and efforts will be made to standardize therapy as much as possible. The evaluating therapist who is blinded to treatment assignment will complete the Fugl-Meyer upper extremity subsection every 6 weeks and the FIM at week 1 and at the final visit. Participants will be seen every 6 weeks by the coordinator and physician for Study Visits 2, 3/3A, 4, and 5 at which time they will have the following assessments: Modified Ashworth Scale (MAS), , Patients' Disability and Carer Burden Rating Scale, Visual Analog Scale and the Disability Assessment Scale. The participants in Cohort 2 will follow the same injection and assessment schedule (including Fugl-Meyer upper extremity subsection every 6 weeks and FIM at week 1 and at the final visit), but will not participate in therapy. If, by visit 3, the participants' upper limb spasticity has reached a MAS score of 2 or greater in the wrist and/or fingers, they will be eligible for a second injection of BoNT-A. Any subjects who do not meet re-injection criteria by Visit 3 (week 12) will be re-evaluated in another 3 weeks, Visit 3A. If participants do not meet re-injection criteria by Study Visit 3A (week 15) they will not receive another injection, but will be followed until Visit 5 (final visit). If subjects are injected at visit 3A, visit 4 will occur at 21 weeks (6 weeks after 2nd injection). Visit 5 will occur at week 27 (12 weeks after 2nd injection). Participants receiving both injections will complete the study no sooner than Study Visit 5. The expected time to recruit patients and complete the study is 18 months.

All participants will be queried at each visit regarding the occurrence of adverse events (AE) or serious adverse events (SAE). All unexpected AE and all SAEs will be reviewed by the Site Principal Investigator and reported to the local IRB and reported to Dr. Glenn Graham who will then report to the VA Research & Development Committee and the University of New Mexico Health Science Center Human Research Review Committee. (See Appendix I for AE and SAE definitions). Study sites will be in regular contact with study participants whether or not they receive weekly therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Stroke (ischemic or hemorrhagic) diagnosed by a neurologist at least 6 months prior to enrollment
* Focal spasticity in upper limb measured at the elbow, wrist, fingers and thumb with a Modified Ashworth Scale (MAS) of 3 or greater in the wrist and/or fingers
* Functional impairment secondary to spasticity such as difficulty with hygiene, dressing, posture or pain
* Minimum weight of 44 kg (88 lbs) in order to tolerate the minimum required dosage of 200 U
* Written informed consent has been obtained
* Written authorization for Use and Release of Health and Research Study Information has been obtained
* Laboratory findings required (if applicable)
* Ability to follow study instructions and likely to complete all required visits
* Negative urine pregnancy test on the day of treatment prior to the administration of study medication (for females of childbearing potential). (If applicable.)

Exclusion Criteria:

* Uncontrolled clinically significant medical condition other than the condition under evaluation
* Known allergy or sensitivity to any of the components in the study medication
* Females who are pregnant, breast-feeding, or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study
* Concurrent participation in another investigational drug or device study or participation in the 30 days immediately prior to study enrollment
* Fixed contracture or profound atrophy in the spastic limb
* Prior or current treatment with neurolytic agents such as phenol or surgery; any version of botulinum toxin (other than BoNT-A more than 6 months prior to enrollment)
* Current rehabilitation therapy that cannot be altered to the treatment plan in the study
* Unable or unwilling to participate in a weekly rehab program
* Any medical condition that may put the subject at increased risk with exposure to BOTOX including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function
* Current treatment with agents affecting neuromuscular transmission
* Evidence of recent alcohol or drug abuse
* Infection or skin disorder at an anticipated injection site (if applicable)
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D. Graham, MD, PhD, Principal Investigator — New Mexico VA Healthcare System
Locations (1):
- New Mexico VA Health Care System, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty one patients with post-stroke upper limb spasticity aged 36 - 75 years were enrolled. Patients were recruited from neurology clinics and through local advertisements.
Pre-assignment Details: At the time of consent, all participants agreed that if they were assigned to the BoNT-A no rehab, they would not to start any new therapy or exercise program for arm spasticity until they were finished with the study.
Groups:
- Cohort #1: Cohort 1 will receive BoNT-A plus rehabilitation therapy for the duration of the study (for up to 2 injections of BoNT-A).
  Rehabilitation Therapy : Rehabilitation therapy
  Botulinum toxin type A, BoNT-A : Participants will receive IM injections of BoNT-A between 200 and 400 Units with the total dose not to exceed 6 U / kg. The primary targets for BoNT-A injection are the wrist and finger flexor muscles (flexor carpi radialis, flexor carpi ulnaris, flexor digitorum profundus, flexor digitorum superficialis).
- Cohort #2: Cohort 2 will receive BoNT-A alone
  Botulinum toxin type A, BoNT-A : Participants will receive IM injections of BoNT-A between 200 and 400 Units with the total dose not to exceed 6 U / kg. The primary targets for BoNT-A injection are the wrist and finger flexor muscles (flexor carpi radialis, flexor carpi ulnaris, flexor digitorum profundus, flexor digitorum superficialis).
Period: Overall Study
Arm/Group | Cohort #1 | Cohort #2
Started | 15 | 16
Completed | 15 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort #1 | Cohort #2 | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 20
  >=65 years | 4 | 7 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.6) | 60.9 (11.0) | 59.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Change in Fugl-Meyer Upper Extremity Score From the Baseline Exam to Any Post Injection Visit in Each Treatment Arm. Comparison of the Difference Scores Between the Two Groups Will be Considered Significant at p < 0.05.
Time Frame: 6 Weeks
Measure: Number; unit: difference
Arm/Group | Cohort #1 | Cohort #2
Number analyzed (Participants) | 15 | 16
difference | 6.86 | 3.55

2. Secondary Outcome: Length of Time to Meet Re-injection Criteria and the Number of Participants That do Not Meet Re-injection Criteria Prior to Completion of the Study.
Time Frame: 6 Weeks
Measure: Number; unit: number
Arm/Group | Cohort #1 | Cohort #2
Number analyzed (Participants) | 15 | 16
number | 4 | 1

ADVERSE EVENTS:
Arm/Group | Cohort #1 | Cohort #2
Serious Adverse Events (participants affected / at risk) | 3/15 | 2/16
Other Adverse Events (participants affected / at risk) | 10/15 | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort #1 (N=15) | Cohort #2 (N=16)
hospitalization (Nervous system disorders) | 3 (3) | 2 (2) — In cohort 1: 1 with a h/o seizures was hospitalized with seizures. 1 fell and hit head. 1 developed an infection within the pocket containing a defibrillator. In cohort 2: 1 participant was hospitalized with food poisoning. 1 fell and broke wrist.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort #1 (N=15) | Cohort #2 (N=16)
seizures (Nervous system disorders) | 2 (2) | 0 (0)
infection (Infections and infestations) | 6 (6) | 2 (2) — Cohort 1: 3 UTIs; 1 cold; 1 pneumonia; 1 infected toe Cohort 2: 2 UTIs
anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Cohort 1: 2 participants with anemia
pain (General disorders) | 0 (0) | 2 (2) — Cohort 2: 1 participant with neck pain; 1 with throat pain

LIMITATIONS AND CAVEATS:
This has a single-blind design. Admittedly, a double-blind design is best, but the participants could not be blind to the assignment of rehabilitation. Secondly, the study involved a relatively small sample size and limited follow-up duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No